CLINICAL TRIAL: NCT02158806
Title: Low Dose Aspirin for Venous Leg Ulcers: a Randomised Trial
Brief Title: Low Dose Aspirin for Venous Leg Ulcers
Acronym: Aspirin4VLU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew Jull, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aspirin4VLU
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Venous Leg Ulcer
Keywords: Venous ulcer, varicose ulcer, gravitational ulcer, aspirin
MeSH Terms: conditions — Varicose Ulcer | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo with only difference being unique code on bottle containing product.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): 150 mg capsule once daily for up to 24 weeks
  Interventions: Drug: Aspirin
- Inert capsule (Placebo Comparator): Matching capsule once daily for up to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 150 mg aspirin in capsule form once daily for up to 24 weeks
  Arms: Aspirin
Drug: Placebo — Matching placebo capsule containing inert bulking agent
  Arms: Inert capsule

SUMMARY:
Venous leg ulcers (VLU) are the most common leg ulcer, can be painful, and limit work, lifestyles and activity, especially in older patients. There are few effective treatments - compression therapy (tight bandaging or stockings) helps healing, but about half the people with a VLU remain unhealed even after 12 weeks of treatment. Research suggests taking aspirin as well as using compression may speed up healing for VLU, but the current evidence is not enough to change clinical practice. We will conduct a randomised controlled trial to test whether using low dose aspirin (150 mg daily or placebo) really does speed up healing.

DETAILED DESCRIPTION:
A pragmatic, community based, double-blind, placebo-controlled, randomised trial to determine whether low dose aspirin accelerates venous leg ulcer healing at 24 weeks when used in addition to compression. Participants in have compression therapy (system of choice guided by patient and/or clinical preference) as delivered through district nursing services at the study centres as a background treatment. Low dose aspirin (150 mg) or placebo will be taken once daily as an oral capsule.

Participants will be district nursing service patients in five study centres in New Zealand with prevalent or incident venous leg ulcers. A venous leg ulcer will be defined as a wound on the lower leg that has remained unhealed for 4 or more weeks, appears to be primarily venous in aetiology with other causative diseases ruled out. If the participant has two or more venous leg ulcers, the largest ulcer will be the reference ulcer.

Participants will receive three visits from the research nurse - visit 1 to screen for eligibility, visit 2 to consent and randomise the participant, visit 3 to collect outcome data. District nurses will continue to visit the participant (about weekly or more frequently if required) to provide routine care between research nurse visits.

Block randomisation will be used, stratified by study centre and prognostic index (ulcer size greater than 5cm2 and ulcer duration greater than 6 months) to ensure a balance of participants within study centres and for participants likely to be slow healers. Research nurses in the study centres will contact a central telephone answering service, provide information on inclusion criteria, exclusion criteria, and relevant clinical history on consented participants. Randomised participants will receive a bottle of 168 capsules of study medication identified only by unique code and will take the capsule until the reference ulcer heals or up to 24 weeks, whichever occurs sooner.

Participants will take the study medication for up to 24 weeks or until the reference ulcer heals. If the participant has a serious adverse event, needs to start taking aspirin, or must stop taking aspirin to use other medications, they will be withdrawn from treatment, although they will still be followed up at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Determined to have a venous leg ulcer (clinical indications of venous ulceration, Ankle Brachial Index ≥ 0.8, and other causative aetiologies ruled out)
* Able to tolerate compression therapy
* Able to provide written informed consent
* Confirmation with participant's general practitioner that the participant can take low dose aspirin or placebo.

Exclusion Criteria:

* Pregnant or breast-feeding women
* History of myocardial infarction, stroke, transient ischaemic attack, angina or significant peripheral arterial disease
* History of adverse effects related to aspirin use
* Currently using aspirin, or other anti-platelet or anticoagulant therapy
* Opinion of screening medical practitioner at National Institute of Health Innovation that participant has an existing condition or treatment that is a contraindication to use of aspirin or to participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Jull, RN PhD, Principal Investigator — School of Nursing, University of Auckland

IPD SHARING:
Plan to Share IPD: Yes
We have a plan to share individual participant data with other aspirin for VLU triallists. All other requests for de-identified individual participant data or study documents will be considered where the proposed use aligns with public good purposes, does not conflict with other requests, or planned use by the Trial Steering Committee, and the requestor is willing to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No limitations to timeframe
Access Criteria: We have a plan to share individual participant data with other aspirin for VLU triallists. All other requests for de-identified individual participant data or study documents will be considered where the proposed use aligns with public good purposes, does not conflict with other requests, or planned use by the Trial Steering Committee, and the requestor is willing to sign a data access agreement.

REFERENCES:
- [Background] Jull A, Wadham A, Bullen C, Parag V, Kerse N, Waters J. Low-dose aspirin as an adjuvant treatment for venous leg ulceration: study protocol for a randomized controlled trial (Aspirin4VLU). J Adv Nurs. 2016 Mar;72(3):669-79. doi: 10.1111/jan.12864. Epub 2015 Dec 28. PMID 26708314
- [Derived] Jull A, Wadham A, Bullen C, Parag V, Kerse N, Waters J. Low dose aspirin as adjuvant treatment for venous leg ulceration: pragmatic, randomised, double blind, placebo controlled trial (Aspirin4VLU). BMJ. 2017 Nov 24;359:j5157. doi: 10.1136/bmj.j5157. PMID 29175902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and recruited from five study sites in New Zealand
Pre-assignment Details: Enrolled participants were required to have their family physician confirm they could safely participate in the trial ie had no conditions that required treatment with aspirin and no conditions that contraindicated use of aspirin.
Groups:
- Placebo: Matching inert capsule once daily for up to 24 weeks
  Placebo: Matching placebo capsule containing inert bulking agent
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 125 | 126
Completed | 121 (We had information on all participants for the primary outcome (time to complete healing).) | 121 (We had information on all participants for the primary outcome (time to complete healing).)
Not Completed | 4 | 5
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Moved out of area | 0 | 1
Not completed — Transferred to palliative care | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (17.1) | 56.2 (16.1) | 58.2 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 65 | 68 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Māori | 21 | 16 | 37
  Pasifika | 23 | 30 | 53
  Asian | 4 | 5 | 9
  NZ European/Pākehā | 77 | 74 | 151
  Other | 0 | 1 | 1
Highest educational attainment [Count of Participants; unit: Participants]
  Primary school | 9 | 6 | 15
  Secondary school | 66 | 74 | 140
  Undergraduate | 9 | 17 | 26
  Postgraduate | 21 | 11 | 32
  Vocational/technical | 20 | 17 | 37
  None | 0 | 1 | 1
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 62 | 63 | 125
  Former smoker | 47 | 44 | 91
  Current smoker | 16 | 19 | 35
Medical history [Count of Participants; unit: Participants]
  Diabetes | 13 | 13 | 26
  Prior DVT | 11 | 7 | 18
  Lower limb joint replacement | 16 | 19 | 35
  Prior lower limb fracture | 18 | 23 | 41
  Prior treatment for varicosities | 35 | 33 | 68
Ankle Brachial Index [Mean (Standard Deviation); unit: Ratio of SBP ankle/SBP arm] | 1.1 (0.1) | 1.1 (0.1) | 1.1 (0.1)
Reference ulcer area [Median (Inter-Quartile Range); unit: square centimetres] | 2.6 [0.9 to 6.8] | 2.3 [0.9 to 6.1] | 2.5 [0.9 to 6.3]
Compression system [Count of Participants; unit: Participants]
  High compression | 105 | 102 | 207
  Light compression | 11 | 11 | 22
  Hosiery | 8 | 13 | 21
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Healing of Reference Ulcer
Description: Time to event (complete healing defined as intact skin with absence of scab)
Time Frame: 24 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 125 | 126
days | 77 [56 to 98] | 69 [56 to 98]
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Placebo group = reference group; Test type: Superiority — Participants analysed in the groups to which they were randomised (intention to treat analysis); p = 0.246, Log Rank; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.64 to 1.13], Standard Error of Mean 0.146 — Placebo group = reference group

2. Secondary Outcome: Number of Participants With Healed Venous Leg Ulcers
Description: Number of participants in each arm with completely healed reference ulcers at 24 weeks
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 125 | 126
Participants | 88 | 101
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority — Participants analysed in the groups to which they were randomised (intention to treat analysis); p = 0.073, Chi-squared; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.76 to 1.01]

3. Secondary Outcome: Change in Estimated Ulcer Area
Description: Change in estimated ulcer area from baseline to 24 weeks
Time Frame: Baseline, 24 weeks
Population: Ulcer area estimated using maximum width and length of the ulcer to calculate the area of an ellipse. We have previously shown this approach to be highly correlated with digital calculation of measured area (r=0.92).
Measure: Mean (Standard Error); unit: square centimetres
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 125 | 126
square centimetres | 4.1 (0.4) | 4.8 (0.4)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority; p = 0.25, ANCOVA — Adjusted for baseline values; One participant in aspirin group had missing data for 24 week endpoint visit; we used the baseline value for imputation; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.9 to 0.5], Standard Error of Mean 0.6 — Placebo group = reference group

4. Secondary Outcome: Change in Health-related Quality of Life (Short Form 36)
Description: Mean difference in change in Short Form 36 (SF36) from baseline to 24 weeks. Crude subscale scores for each group are not shown (each crude subscale is scored 0 to 100 at baseline and 24 weeks); higher mean differences in change from baseline to 24 weeks within groups indicate greater change on the subscales for that group.
Time Frame: Baseline, 24 weeks
Population: Only participants that provided both baseline and endpoint data were included in the analysis. Hence the number of participants included in this analysis is less than the number randomized.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 116 | 115
units on a scale
  Physical Functioning | 5.0 (2.2) | 3.8 (2.2)
  Role Physical | 11.7 (3.4) | 10.3 (3.4)
  Bodily Pain | 11.4 (2.2) | 9.0 (2.2)
  General Health | -1.1 (1.4) | -0.8 (1.4)
  Vitality | 3.9 (1.6) | -0.3 (1.6)
  Social Functioning | 5.8 (2.2) | 4.9 (2.2)
  Role Emotional | 10.5 (3.1) | 6.8 (3.1)
  Mental Health | -1.2 (1.4) | 1.2 (1.4)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Change in Physical Functioning; Test type: Superiority; p = 0.714, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 1.1, 95% CI 2-sided [-5.0 to 7.2]
Statistical Analysis 2: Comparison: Aspirin vs Placebo; Change in Role Physical; Test type: Superiority; p = 0.768, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 1.4, 95% CI 2-sided [-8.0 to 10.8]
Statistical Analysis 3: Comparison: Aspirin vs Placebo; Change in Bodily Pain; Test type: Superiority; p = 0.449, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 2.3, 95% CI 2-sided [-3.7 to 8.4]
Statistical Analysis 4: Comparison: Aspirin vs Placebo; Change in General Health; Test type: Superiority; p = 0.873, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -0.3, 95% CI 2-sided [-4.3 to 3.6]
Statistical Analysis 5: Comparison: Aspirin vs Placebo; Change in Vitality; Test type: Superiority; p = 0.057, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 4.2, 95% CI 2-sided [-0.1 to 8.5]
Statistical Analysis 6: Comparison: Aspirin vs Placebo; Change in Social Functioning; Test type: Superiority; p = 0.756, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 1.0, 95% CI 2-sided [-5.1 to 7.0]
Statistical Analysis 7: Comparison: Aspirin vs Placebo; Change in Role Emotional; Test type: Superiority; p = 0.400, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 3.7, 95% CI 2-sided [-4.9 to 12.3]
Statistical Analysis 8: Comparison: Aspirin vs Placebo; Change in Mental Health; Test type: Superiority; p = 0.236, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -2.3, 95% CI 2-sided [-6.2 to 1.5]

5. Secondary Outcome: Change in Health-related Quality of Life (EuroQol-5D 3L)
Description: Mean difference in change measured by EuroQol 5D (EQ5D 3L) from baseline to 24 weeks. Crude health state scores for each group are not shown (health state is scored 0 to 100 at baseline and 24 weeks); higher mean differences in change from baseline to 24 weeks within groups indicate greater change on health state for that group.
Time Frame: Baseline, 24 weeks
Population: Only participants that provided both baseline and endpoint data were included in the analysis. Hence the number of participants included in this analysis is less than the number randomised.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 116 | 115
score on a scale | 7.4 (1.6) | 4.0 (1.7)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority; p = 0.156, Regression, Linear — Adjusted for baseline values; Mean Difference (Net) = 3.4, 95% CI 2-sided [-1.3 to 8.0]

6. Secondary Outcome: Change in Health-related Quality of Life (Charing Cross Venous Ulcer Questionnaire)
Description: Mean difference in change in Charing Cross Venous Ulcer Questionnaire (CXVUQ)) from baseline to 24 weeks. Crude subscale scores for each group are not shown (each crude subscale is scored 0 to 100 at baseline and 24 weeks); higher mean differences in change from baseline to 24 weeks within groups indicate greater change on the subscales for that group.
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 115 | 116
score on a scale
  Social function | -6.2 (1.3) | -4.7 (1.3)
  Domestic activities | -6.6 (1.1) | -5.2 (1.2)
  Cosmesis | -6.1 (1.6) | -4.9 (1.6)
  Emotional status | -9.4 (1.8) | -6.5 (1.8)
  Overall | -7.3 (1.2) | -5.5 (1.2)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Change in social function; Test type: Superiority; p = 0.438, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -1.5, 95% CI 2-sided [-5.2 to 2.2]
Statistical Analysis 2: Comparison: Aspirin vs Placebo; Change in domestic activities; Test type: Superiority; p = 0.408, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -1.3, 95% CI 2-sided [-4.5 to 1.9]
Statistical Analysis 3: Comparison: Aspirin vs Placebo; Change in cosmesis; Test type: Superiority; p = 0.568, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -1.3, 95% CI 2-sided [-5.6 to 3.1]
Statistical Analysis 4: Comparison: Aspirin vs Placebo; Change in emotional status; Test type: Superiority; p = 0.257, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -3.0, 95% CI 2-sided [-8.1 to 2.2]
Statistical Analysis 5: Comparison: Aspirin vs Placebo; Test type: Superiority; p = 0.273, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -1.9, 95% CI 2-sided [-5.2 to 1.5]

7. Secondary Outcome: Number of Participants With Adherence to Treatment
Description: Adherence to study medication as measured by pill counts (agreement between expected number of tablets remaining after healing and days to healing)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 125 | 126
Participants | 92 | 92
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority; p = 0.917, Chi-squared; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.87 to 1.17]

8. Secondary Outcome: Incidence of Adverse Events at 24 Weeks
Description: Total number of different types of adverse events in participants who reported with any untoward medical event
Time Frame: 24 weeks
Population: Only participants that reported any reported untoward medical event were included in this analysis.
Measure: Count of Units; unit: Number of events
Units Other Than Participants: Number of events
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 29 | 27
Number analyzed (Number of events) | 40 | 37
Number of events
  Cancer | 6 | 1
  Cardiovascular | 0 | 4
  Gastrointestinal | 8 | 4
  Respiratory | 3 | 0
  Genitourinary | 2 | 0
  Skin & cutaneous | 1 | 5
  Accidental injury | 4 | 4
  Psychiatric | 1 | 0
  Signs & symptoms | 7 | 5
  Leg ulcer bleeding | 2 | 2
  Leg ulcer infection | 2 | 4
  Extension of leg ulcer | 1 | 2
  New leg ulcer | 1 | 3
  Other | 2 | 3
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority; p = 0.71, IRR test statistic; Incidence Rate Ratio (IRR) test statistic compared to probability of the same obtained from standard normal distribution tables; Incidence Rate Ratio = 1.1, 95% CI 2-sided [0.7 to 1.7]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Aspirin | Placebo
All-Cause Mortality (participants affected / at risk) | 2/125 | 0/126
Serious Adverse Events (participants affected / at risk) | 11/125 | 10/126
Other Adverse Events (participants affected / at risk) | 20/125 | 18/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=125) | Placebo (N=126)
Hospitalisation or prolongation of hospitalisation (Infections and infestations) | 0 (0) | 1 (1) — Staphylococcal infection, unspecified site
Hospitalisation or prolongation of hospitalisation (Infections and infestations) | 1 (1) | 0 (0) — Infection of ulceration
Hospitalisation or prolongation of hospitalisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) — Metastatic squamous cell carcinoma
Hospitalisation or prolongation of hospitalisation (Cardiac disorders) | 0 (0) | 1 (1) — Other cardiomyopathies
Hospitalisation or prolongation of hospitalisation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Phlebitis and thrombophlebitis of other deep vessels of lower extremities
Hospitalisation or prolongation of hospitalisation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumonitis due to food and vomit
Hospitalisation or prolongation of hospitalisation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Volvulus
Hospitalisation or prolongation of hospitalisation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Constipation
Hospitalisation or prolongation of hospitalisation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Haemorrhage of anus and rectum
Hospitalisation or prolongation of hospitalisation (Gastrointestinal disorders) | 1 (1) | 1 (1) — Gastrointestinal haemorrhage, unspecified
Hospitalisation or prolongation of hospitalisation (Infections and infestations) | 1 (1) | 3 (3) — Cellulitis of lower limb
Hospitalisation or prolongation of hospitalisation (Renal and urinary disorders) | 1 (1) | 0 (0) — Acute kidney failure, unspecified
Hospitalisation or prolongation of hospitalisation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Pharyngeal pouch
Hospitalisation or prolongation of hospitalisation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Epistaxis
Hospitalisation or prolongation of hospitalisation (Cardiac disorders) | 1 (1) | 0 (0) — Chest pain, unspecified
Hospitalisation or prolongation of hospitalisation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Other and unspecified abdominal pain
Hospitalisation or prolongation of hospitalisation (Cardiac disorders) | 0 (0) | 1 (1) — Syncope and collapse
Hospitalisation or prolongation of hospitalisation (General disorders) | 1 (2) | 0 (0) — Malaise and fatigue
Hospitalisation or prolongation of hospitalisation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Fracture shaft of tibia with fracture of fibula (any part)
Hospitalisation or prolongation of hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0) — Presence of hip implant
Life threatening event of illness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Malignant neoplasm of brain, unspecified
Significan medical event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) — Malignant neoplasm of breast, unspecified part
Significant medical event (Immune system disorders) | 0 (0) | 1 (1) — Allergy, unspecified
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Malignant neoplasm of prostate
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Other unspecified respiratory disorder
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=125) | Placebo (N=126)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Other specified respiratory disorders
Bleeding from any lower leg ulceration (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Infection of ulceration, any lower leg ulceration (Infections and infestations) | 1 (1) | 3 (4)
Developed any new lower leg ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Extension of reference ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — Including incorporation of other ulcers into reference ulcer
Candidal stomatitis (Infections and infestations) | 0 (0) | 1 (1)
Coagulation defect, unspecified (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Longer bleeding time on small cuts to hands
Depressive episode, unspecified (Psychiatric disorders) | 1 (1) | 0 (0)
Acute inflammation of orbit (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Varicose veins of lower extremities with inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Varicose veins of lower extremities without ulcer or inflammation (Vascular disorders) | 0 (0) | 1 (1) — Saphenous femoral junction incompetence, other leg
Gastro-oesophageal reflux disease without oesophagi's (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer, unspecified as acute or chronic, without haemorrhage or perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis, unspecified (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis of lower limb (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urinary tract infection, site not specified (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Tendency to fall, not elsewhere classified (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperhidrosis (General disorders) | 0 (0) | 1 (1)
Laceration and contusions (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Allergy, unspecified (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was lower than anticipated as fewer aspirin-naive patients being available than estimated. However we had 82% power to observe the anticipated difference if assumptions had been correct.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-05-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT02158806/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT02158806/SAP_001.pdf
  • Informed Consent Form (2014-08-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT02158806/ICF_002.pdf